CLINICAL TRIAL: NCT03187418
Title: Treatment Outcomes of MicroPulse Trans-scleral Cyclophotocoagulation (mTSCPC) in Uncontrolled Glaucoma at the University of Montreal Hospital Center (CHUM)
Brief Title: Treatment Outcomes of MicroPulse Trans-scleral Cyclophotocoagulation in Uncontrolled Glaucoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CE16.351
Record Dates: First submitted 2017-06-12; First posted 2017-06-15 (Actual); Results first posted 2021-10-08 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2020-08

CONDITIONS: Glaucoma; Glaucoma, Open-Angle; Glaucoma, Neovascular; Glaucoma and Ocular Hypertension; Glaucoma Eye; Glaucoma, Uncompensated; Glaucoma Secondary
Keywords: Cyclophotocoagulation; Micropulse TSCPC; Laser ablation; Laser therapy
MeSH Terms: conditions — Glaucoma; Glaucoma, Open-Angle; Glaucoma, Neovascular; Ocular Hypertension; Glaucoma, Angle-Closure

STUDY DESIGN:
Intervention Model Description: Prospective, interventional and monocentric study based in a university hospital setting
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Micropulse trans-scleral CPC (Experimental): A treatment session of micropulse trans-scleral cyclophotocoagulation in the affected eye, using the MicroPulse® P3 Glaucoma Device (MP3) powered by the CYCLO G6™ Glaucoma Laser System (Iridex, Mountain View, CA, USA).
  Interventions: Device: MicroPulse® P3 Glaucoma Device (MP3)

INTERVENTIONS:
Device: MicroPulse® P3 Glaucoma Device (MP3) — Laser settings will be programmed as follows: power-2000mW-2500mW (average 2000mW) of 810nm infrared diode laser set on micropulse delivery mode; micropulse "on" time-0.5ms; micropulse "off" time-1.1ms; and duty cycle (proportion of each cycle during which the laser is on)-31.33 %.
  The laser probe will be applied in a continuous sliding or painting motion from 9:30 to 2:30 and from 3:30 to 8:30. The probe will be applied perpendicular to the limbus with the edge directly on the limbus at all times (fiberoptic tip at 3 mm posterior to the limbus).
  The laser will be delivered over 360° for 160-320s. Treatment duration will be adjusted based on iris color and glaucoma severity (mild glaucoma: 160s, moderate glaucoma: 240s, advanced glaucoma: 240-320s).
  Other Names: CYCLO G6 Glaucoma Laser System (Iridex, Mountain View, CA)

SUMMARY:
The goal of this study is to evaluate the efficacy and safety of the novel form of trans-scleral cyclophotocoagulation using micropulse diode laser and trans-pars plana treatment (Micropulse TSCPC, mTSCPC MP3, IRIDEX CYCLO G6™ Glaucoma Laser System, CA, USA) in adults for the treatment of uncontrolled glaucoma.

DETAILED DESCRIPTION:
Cyclophotocoagulation (CPC) is a type of cycloablation using laser to treat glaucoma. It involves ciliary body destruction by targeting the ciliary epithelium and stroma, resulting in a reduction in aqueous secretion and hence intraocular pressure. This strategy is effective for all forms of glaucoma.

Traditional trans-scleral cyclophotocoagulation (TSCPC) achieve its cyclodestructive action by using continuous diode laser to target the melanin in the pigmented ciliary body epithelium. However, the continuous mode has been shown to cause significant collateral tissue damage to adjacent non-pigmented structures including the ciliary stroma and ciliary muscle. Traditional TSCPC may therefore be associated with serious complications including uveitis, visual deterioration, chronic hypotony, and others.

More recently, a micropulse delivery mode of diode laser (Micropulse TSCPC, mTSCPC) has been used to treat glaucoma by ablating the ciliary processes and reduce aqueous humor production with more selective targeting and less collateral damage. In contrast to conventional laser delivery where a continuous flow of high intensity energy is delivered, micropulse laser application delivers a series of repetitive short pulses of energy with rest periods in between pulses. Only a few studies have described the outcomes of this novel glaucoma therapy, showing mTSCPC to have comparable efficacy with fewer side effects when compared with traditional continuous wave mode diode laser delivery.This improved side effect profile has the potential to make mTSCPC an earlier therapeutic option instead of reserving it exclusively for end-stage refractory eyes.

ELIGIBILITY:
Inclusion Criteria:

* Patients of either sex and any race aged 18 years old and above.
* Followed by a glaucoma subspecialist at University of Montreal Hospital Center.
* Intraocular pressure (IOP) above target and unresponsive to maximal tolerated medical therapy with or without previous surgical intervention.

  1. mild glaucoma: IOP > 18 mmHg
  2. moderate glaucoma: IOP > 15 mmHg
  3. advanced glaucoma: IOP > 12 mmHg
* Considered poor candidates for additional filtering surgery or implantation of glaucoma drainage devices.

Exclusion Criteria:

* Patients unable to give informed consent.
* Patients with significant scleral thinning, defined as thinning of more than one clock hour noticed on scleral transillumination.
* Ocular infection or inflammation in the study eye in the 2 months prior to enrolment.
* Intraocular surgery in the study eye in the 2 months prior to enrolment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2017-06-19 (Actual); Primary Completion 2020-02-15 (Actual); Study Completion 2020-02-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harmanjit Singh, MD, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM); Michael Marchand, MD, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Quigley HA, Broman AT. The number of people with glaucoma worldwide in 2010 and 2020. Br J Ophthalmol. 2006 Mar;90(3):262-7. doi: 10.1136/bjo.2005.081224. PMID 16488940
- [Background] Tham YC, Li X, Wong TY, Quigley HA, Aung T, Cheng CY. Global prevalence of glaucoma and projections of glaucoma burden through 2040: a systematic review and meta-analysis. Ophthalmology. 2014 Nov;121(11):2081-90. doi: 10.1016/j.ophtha.2014.05.013. Epub 2014 Jun 26. PMID 24974815
- [Background] Nguyen QH. Primary surgical management refractory glaucoma: tubes as initial surgery. Curr Opin Ophthalmol. 2009 Mar;20(2):122-5. doi: 10.1097/ICU.0b013e32831da828. PMID 19240544
- [Background] Schlote T, Derse M, Rassmann K, Nicaeus T, Dietz K, Thiel HJ. Efficacy and safety of contact transscleral diode laser cyclophotocoagulation for advanced glaucoma. J Glaucoma. 2001 Aug;10(4):294-301. doi: 10.1097/00061198-200108000-00009. PMID 11558814
- [Background] Agarwal HC, Gupta V, Sihota R. Evaluation of contact versus non-contact diode laser cyclophotocoagulation for refractory glaucomas using similar energy settings. Clin Exp Ophthalmol. 2004 Feb;32(1):33-8. doi: 10.1046/j.1442-9071.2004.00754.x. PMID 14746588
- [Background] Schlote T, Derse M, Zierhut M. Transscleral diode laser cyclophotocoagulation for the treatment of refractory glaucoma secondary to inflammatory eye diseases. Br J Ophthalmol. 2000 Sep;84(9):999-1003. doi: 10.1136/bjo.84.9.999. PMID 10966953
- [Background] Egbert PR, Fiadoyor S, Budenz DL, Dadzie P, Byrd S. Diode laser transscleral cyclophotocoagulation as a primary surgical treatment for primary open-angle glaucoma. Arch Ophthalmol. 2001 Mar;119(3):345-50. doi: 10.1001/archopht.119.3.345. PMID 11231767
- [Background] Leszczynski R, Gierek-Lapinska A, Forminska - Kapuscik M. Transscleral cyclophotocoagulation in the treatment of secondary glaucoma. Med Sci Monit. 2004 Sep;10(9):CR542-8. Epub 2004 Aug 20. PMID 15328489
- [Background] Rotchford AP, Jayasawal R, Madhusudhan S, Ho S, King AJ, Vernon SA. Transscleral diode laser cycloablation in patients with good vision. Br J Ophthalmol. 2010 Sep;94(9):1180-3. doi: 10.1136/bjo.2008.145565. Epub 2010 Jun 24. PMID 20576775
- [Background] Pantcheva MB, Kahook MY, Schuman JS, Rubin MW, Noecker RJ. Comparison of acute structural and histopathological changes of the porcine ciliary processes after endoscopic cyclophotocoagulation and transscleral cyclophotocoagulation. Clin Exp Ophthalmol. 2007 Apr;35(3):270-4. doi: 10.1111/j.1442-9071.2006.01415.x. PMID 17430515
- [Background] Tan AM, Chockalingam M, Aquino MC, Lim ZI, See JL, Chew PT. Micropulse transscleral diode laser cyclophotocoagulation in the treatment of refractory glaucoma. Clin Exp Ophthalmol. 2010 Apr;38(3):266-72. doi: 10.1111/j.1442-9071.2010.02238.x. PMID 20447122
- [Background] Aquino MC, Barton K, Tan AM, Sng C, Li X, Loon SC, Chew PT. Micropulse versus continuous wave transscleral diode cyclophotocoagulation in refractory glaucoma: a randomized exploratory study. Clin Exp Ophthalmol. 2015 Jan-Feb;43(1):40-6. doi: 10.1111/ceo.12360. Epub 2014 Jun 21. PMID 24811050
- [Background] Bloom PA, Tsai JC, Sharma K, Miller MH, Rice NS, Hitchings RA, Khaw PT. "Cyclodiode". Trans-scleral diode laser cyclophotocoagulation in the treatment of advanced refractory glaucoma. Ophthalmology. 1997 Sep;104(9):1508-19; discussion 1519-20. doi: 10.1016/s0161-6420(97)30109-2. PMID 9307649
- [Background] Kosoko O, Gaasterland DE, Pollack IP, Enger CL. Long-term outcome of initial ciliary ablation with contact diode laser transscleral cyclophotocoagulation for severe glaucoma. The Diode Laser Ciliary Ablation Study Group. Ophthalmology. 1996 Aug;103(8):1294-302. doi: 10.1016/s0161-6420(96)30508-3. PMID 8764801
- [Background] Mistlberger A, Liebmann JM, Tschiderer H, Ritch R, Ruckhofer J, Grabner G. Diode laser transscleral cyclophotocoagulation for refractory glaucoma. J Glaucoma. 2001 Aug;10(4):288-93. doi: 10.1097/00061198-200108000-00008. PMID 11558813
- [Background] Oguri A, Takahashi E, Tomita G, Yamamoto T, Jikihara S, Kitazawa Y. Transscleral cyclophotocoagulation with the diode laser for neovascular glaucoma. Ophthalmic Surg Lasers. 1998 Sep;29(9):722-7. PMID 9760607
- [Background] Sivaprasad S, Sandhu R, Tandon A, Sayed-Ahmed K, McHugh DA. Subthreshold micropulse diode laser photocoagulation for clinically significant diabetic macular oedema: a three-year follow up. Clin Exp Ophthalmol. 2007 Sep-Oct;35(7):640-4. doi: 10.1111/j.1442-9071.2007.01566.x. PMID 17894684
- [Background] Parodi MB, Spasse S, Iacono P, Di Stefano G, Canziani T, Ravalico G. Subthreshold grid laser treatment of macular edema secondary to branch retinal vein occlusion with micropulse infrared (810 nanometer) diode laser. Ophthalmology. 2006 Dec;113(12):2237-42. doi: 10.1016/j.ophtha.2006.05.056. Epub 2006 Sep 25. PMID 16996596
- [Background] Desmettre TJ, Mordon SR, Buzawa DM, Mainster MA. Micropulse and continuous wave diode retinal photocoagulation: visible and subvisible lesion parameters. Br J Ophthalmol. 2006 Jun;90(6):709-12. doi: 10.1136/bjo.2005.086942. Epub 2006 Mar 10. PMID 16531424
- [Background] Laursen ML, Moeller F, Sander B, Sjoelie AK. Subthreshold micropulse diode laser treatment in diabetic macular oedema. Br J Ophthalmol. 2004 Sep;88(9):1173-9. doi: 10.1136/bjo.2003.040949. PMID 15317711
- [Background] Moorman CM, Hamilton AM. Clinical applications of the MicroPulse diode laser. Eye (Lond). 1999 Apr;13 ( Pt 2):145-50. doi: 10.1038/eye.1999.41. PMID 10450372
- [Background] Pollack JS, Kim JE, Pulido JS, Burke JM. Tissue effects of subclinical diode laser treatment of the retina. Arch Ophthalmol. 1998 Dec;116(12):1633-9. doi: 10.1001/archopht.116.12.1633. PMID 9869794
- [Background] Berger JW. Thermal modelling of micropulsed diode laser retinal photocoagulation. Lasers Surg Med. 1997;20(4):409-15. doi: 10.1002/(sici)1096-9101(1997)20:43.0.co;2-u. PMID 9142680
- [Background] Kuchar S, Moster MR, Reamer CB, Waisbourd M. Treatment outcomes of micropulse transscleral cyclophotocoagulation in advanced glaucoma. Lasers Med Sci. 2016 Feb;31(2):393-6. doi: 10.1007/s10103-015-1856-9. Epub 2015 Dec 29. PMID 26714976
- [Background] Hauber FA, Scherer WJ. Influence of total energy delivery on success rate after contact diode laser transscleral cyclophotocoagulation: a retrospective case review and meta-analysis. J Glaucoma. 2002 Aug;11(4):329-33. doi: 10.1097/00061198-200208000-00009. PMID 12169970
- [Background] Vernon SA, Koppens JM, Menon GJ, Negi AK. Diode laser cycloablation in adult glaucoma: long-term results of a standard protocol and review of current literature. Clin Exp Ophthalmol. 2006 Jul;34(5):411-20. doi: 10.1111/j.1442-9071.2006.01241.x. PMID 16872335
- [Background] Murphy CC, Burnett CA, Spry PG, Broadway DC, Diamond JP. A two centre study of the dose-response relation for transscleral diode laser cyclophotocoagulation in refractory glaucoma. Br J Ophthalmol. 2003 Oct;87(10):1252-7. doi: 10.1136/bjo.87.10.1252. PMID 14507761
- [Background] Meyer JJ, Lawrence SD. What's new in laser treatment for glaucoma? Curr Opin Ophthalmol. 2012 Mar;23(2):111-7. doi: 10.1097/ICU.0b013e32834f1887. PMID 22186007
- [Derived] Marchand M, Singh H, Agoumi Y. Micropulse trans-scleral laser therapy outcomes for uncontrolled glaucoma: a prospective 18-month study. Can J Ophthalmol. 2021 Dec;56(6):371-378. doi: 10.1016/j.jcjo.2021.01.015. Epub 2021 Feb 10. PMID 33577756

RESULTS

PARTICIPANT FLOW:
Groups:
- Micropulse Trans-scleral CPC: A treatment session of micropulse trans-scleral cyclophotocoagulation in the affected eye, using the MicroPulse® P3 Glaucoma Device (MP3) powered by the CYCLO G6™ Glaucoma Laser System (Iridex, Mountain View, CA, USA).
  MicroPulse® P3 Glaucoma Device (MP3): Laser settings will be programmed as follows: power-2000mW-2500mW (average 2000mW) of 810nm infrared diode laser set on micropulse delivery mode; micropulse "on" time-0.5ms; micropulse "off" time-1.1ms; and duty cycle (proportion of each cycle during which the laser is on)-31.33 %.
  The laser probe will be applied in a continuous sliding or painting motion from 9:30 to 2:30 and from 3:30 to 8:30. The probe will be applied perpendicular to the limbus with the edge directly on the limbus at all times (fiberoptic tip at 3 mm posterior to the limbus).
  The laser will be delivered over 360° for 160-320s. Treatment duration will be adjusted based on iris color and glaucoma severity (mild glaucoma: 160s, moderate glaucoma: 240s, advanced glaucoma: 240-320s).
Period: Overall Study
Arm/Group | Micropulse Trans-scleral CPC
Started | 52
Completed | 52
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Micropulse Trans-scleral CPC
Number analyzed (Participants) | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 69 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 26
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 41
  African American | 6
  Middle East | 3
  Asian | 2
Region of Enrollment [Number; unit: participants]
  Canada | 52
Glaucoma diagnosis [Count of Participants; unit: Participants]
  Primary open angle glaucoma | 28
  Neovascular glaucoma | 5
  Pseudoexfoliative glaucoma | 4
  Congenital/infantile glaucoma | 4
  Chronic primary angle-closure glaucoma | 3
  Pigmentary glaucoma | 3
  Other secondary glaucoma | 2
  Uveitic/inflammatory glaucoma | 1
  Combined mechanism glaucoma | 1
  Normotensive glaucoma | 1
Glaucoma severity [Count of Participants; unit: Participants]
  Mild | 1
  Moderate | 16
  Advanced | 35

OUTCOME MEASURES:

1. Primary Outcome: Intraocular Pressure (IOP)
Description: In millimeters of mercury (mmHg), measured with the Goldmann applanation tonometer
Time Frame: 18 months
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mm Hg)
Arm/Group | Micropulse Trans-scleral CPC
Number analyzed (Participants) | 52
millimeters of mercury (mm Hg) | 15.2 (4.1)

2. Secondary Outcome: Intraocular Pressure (IOP)
Description: In millimeters of mercury (mmHg), measured with the Goldmann applanation tonometer
Time Frame: 1 week, 1 month, 3 months, 6 months, 12 months
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mm Hg)
Arm/Group | Micropulse Trans-scleral CPC
Number analyzed (Participants) | 52
millimeters of mercury (mm Hg)
  1 week | 18.2 (6.3)
  1 month | 19.2 (7.4)
  3 months | 18.6 (6.2)
  6 months | 17.9 (5.3)
  12 months | 16.7 (5.6)

3. Secondary Outcome: Number of Participants With Repeat Treatments
Description: Number of participants needing a repeat laser treatment during the study
Time Frame: 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Micropulse Trans-scleral CPC
Number analyzed (Participants) | 52
Participants | 10

4. Secondary Outcome: Number of Intraocular Pressure Lowering Medications
Description: Number of drops and oral medications used by the patient compared to baseline
Time Frame: 1 week, 1 month, 3 months, 6 months, 12 months, 18 months
Measure: Mean (Standard Deviation); unit: glaucoma medication classes
Arm/Group | Micropulse Trans-scleral CPC
Number analyzed (Participants) | 52
glaucoma medication classes
  1 week | 3.5 (0.7)
  1 month | 3.4 (0.8)
  3 months | 3.4 (0.9)
  6 months | 3.4 (0.8)
  12 months | 3.2 (0.9)
  18 months | 3.2 (0.9)

5. Secondary Outcome: Corrected Distance Visual Acuity (CDVA)
Description: Number of lines reduction or improvement from baseline on Snellen acuity chart at 6 meters
Time Frame: 1 week, 1 month, 3 months, 6 months, 12 months, 18 months
Measure: Mean (Standard Deviation); unit: LogMAR
Arm/Group | Micropulse Trans-scleral CPC
Number analyzed (Participants) | 52
LogMAR
  1 week | 0.81 (0.86)
  1 month | 0.84 (0.90)
  3 months | 0.79 (0.88)
  6 months | 0.77 (0.86)
  12 months | 0.79 (0.86)
  18 months | 0.82 (0.88)

6. Secondary Outcome: Cup-to-disc Ratio (CDR)
Description: Progression of CDR compared to baseline, assessed by an ophthalmologist on dilated fundus examination
Time Frame: 18 months
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Micropulse Trans-scleral CPC
Number analyzed (Participants) | 52
ratio | 0.82 (0.13)

7. Secondary Outcome: Visual Field Index (VFI)
Description: Determined by Humphrey automated perimetry Sita 24-2 visual field testing
Time Frame: 18 months
Measure: Mean (Standard Deviation); unit: percents
Arm/Group | Micropulse Trans-scleral CPC
Number analyzed (Participants) | 52
percents | 57 (27)

8. Secondary Outcome: Mean Deviation (MD)
Description: Determined by Humphrey automated perimetry Sita 24-2 visual field testing
Time Frame: 18 months
Measure: Mean (Standard Deviation); unit: decibel (dB)
Arm/Group | Micropulse Trans-scleral CPC
Number analyzed (Participants) | 52
decibel (dB) | -15.16 (7.72)

9. Secondary Outcome: Pattern Standard Deviation (PSD)
Description: Determined by Humphrey automated perimetry Sita 24-2 visual field testing
Time Frame: 18 months
Measure: Mean (Standard Deviation); unit: decibel (dB)
Arm/Group | Micropulse Trans-scleral CPC
Number analyzed (Participants) | 52
decibel (dB) | 7.87 (3.18)

10. Secondary Outcome: Average Retinal Nerve Fiber Layer (RNFL) Thickness
Description: In micrometer, determined by optical coherence tomography (OCT)
Time Frame: 18 months
Measure: Mean (Standard Deviation); unit: micrometers
Arm/Group | Micropulse Trans-scleral CPC
Number analyzed (Participants) | 52
micrometers | 62 (12)

11. Secondary Outcome: Average Ganglion Cell Layer (GCL) Thickness
Description: In micrometer, determined by optical coherence tomography (OCT)
Time Frame: 18 months
Measure: Mean (Standard Deviation); unit: micrometers
Arm/Group | Micropulse Trans-scleral CPC
Number analyzed (Participants) | 52
micrometers | 53 (14)

12. Secondary Outcome: Cup-to-disc Ratio (CDR) Assessed by Optical Coherence Tomography (OCT)
Description: Progression of vertical CDR compared to baseline, assessed by optical coherence tomography (OCT) parameters
Time Frame: 18 months
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Micropulse Trans-scleral CPC
Number analyzed (Participants) | 52
ratio | 0.82 (0.13)

13. Secondary Outcome: Pain Level During Laser Treatment
Description: Using a verbal analog scale for pain level (none = no subjective feeling of pain, mild = pain easily tolerable, moderate = pain tolerable with difficulty, severe = pain intolerable)
Time Frame: 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | Micropulse Trans-scleral CPC
Number analyzed (Participants) | 52
Participants
  None | 34
  Mild | 12
  Moderate | 6
  Severe | 0

ADVERSE EVENTS:
Time Frame: 18 months
Description: All participants completed the study without any adverse events after 18 months of follow-up. All-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed beyond 18 months.
Arm/Group | Micropulse Trans-scleral CPC
All-Cause Mortality (participants affected / at risk) | 0/52
Serious Adverse Events (participants affected / at risk) | 0/52
Other Adverse Events (participants affected / at risk) | 0/52

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-14): https://cdn.clinicaltrials.gov/large-docs/18/NCT03187418/Prot_SAP_000.pdf